CLINICAL TRIAL: NCT06060483
Title: Effect of Patient Management Based on Continuous Continuous Glucose Monitoring on Major Adverse Cardiovascular Events in Patients With Type 2 Diabetes and Moderate to Severe Coronary Artery Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, zhengchao, Professor Zhengchao, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CGM-MACE
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2; Major Adverse Cardiac Events
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM group (Experimental): Wear CGM continuously and manage patients based on CGM. The treatment goals are TIR>70%, TBR<4%, TAR<25%, and HbA1c<7.0%. After the treatment reaches the standard, CGM is worn every six months.
  Interventions: Device: CGM
- HbA1c group (No Intervention): HbA1c testing is performed every three months, patient management is based on HbA1c, and the treatment target is HbA1c <7.0%.

INTERVENTIONS:
Device: CGM — Wear CGM continuously and manage patients based on CGM. The treatment goals are TIR>70%, TBR<4%, TAR<25%, and HbA1c<7.0%. After the treatment reaches the standard, CGM is worn every six months.
  Arms: CGM group

SUMMARY:
Patients with type 2 diabetes and moderate to severe coronary artery stenosis who were treated at Zhejiang Second Hospital and cooperative hospitals were randomly divided into a patient management group based on continuous continuous glucose monitoring (CGM) or a patient management group based on HbA1c. Both groups controlled cardiovascular risk factors according to the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes (2020) and the ADA Guidelines for the Prevention and Treatment of Diabetes (2023), and conducted HbA1c testing every 3 months. In the CGM-based glucose management group, CGM measurements will be performed at baseline and at 6, 12, 18, and 24 months. In the CGM-guided treatment group, the target TIR>70%, TBR<4%, TAR<25%, and HbA1c<7.0%; in the HbA1c-guided treatment group, the target HbA1c<7.0%. The primary endpoint was major adverse cardiovascular events (MACE: CV death, nonfatal myocardial infarction, nonfatal stroke).

ELIGIBILITY:
Inclusion Criteria:

Male or female between 35 and 75 years old type 2 diabetes HbA1C: 7.5%-10% Moderate to severe coronary artery stenosis (the degree of stenosis of any major coronary artery is ≥50% as assessed by coronary angiography or coronary CTA) The blood sugar lowering regimen has been stable in the past 3 months Ability to understand the requirements of the study and provide informed consent

Exclusion Criteria:

Type 1 diabetes or other types of diabetes Acute myocardial infarction or stroke within the past three months Ketoacidosis, hyperosmolar hyperglycemic state Relative or absolute contraindications to contrast agent examinations such as severe renal insufficiency, contrast agent allergy, and hyperthyroidism Elective surgery planned within 2 years Preparing for pregnancy or becoming pregnant Life expectancy less than 2 years Skin allergies and other situations where CGM cannot be used Currently participating in other clinical studies

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital Zhejiang University Schoolof Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided